CLINICAL TRIAL: NCT06315764
Title: Effect of the Reflexology Versus Aerobic Training on Insomnia Severity Index and Quality of Life in Hypertensive Patients
Brief Title: Effect of the Reflexology on Insomnia Severity Index in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Mousa Galeb, Lecturer at the Department of Physical Therapy for Cardiovascular /Respiratory Disorders and Geriatrics Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hypertensive patients
Record Dates: First submitted 2024-03-05; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
Keywords: Reflexology, Insomina Severity Index; Hypertensive patients.
MeSH Terms: conditions — Hypertension | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Group (A):
  It consists of twenty female patients suffering from hypertension who underwent medical treatment as well as peddler training three times per week for eight weeks. After four weeks of treatment (post-1) and another four weeks of treatment, the post evaluation was used (post-2).
  Group (B):
  This group consisted of twenty female patients suffering from hypertension who received the same drugs as group (A) as well as reflexology three times per week for eight weeks
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic training (Experimental): Each patient in this study did 20 minutes of peddler aerobic training, with the first 5 minutes serving as a warm-up with intensity set at 60 - 65 percent of maximal heart rate, followed by another 10 minutes of peddler training with intensity gradually increased up to 70 - 75 percent, and the last 5 minutes serving as a cooling down with intensity set at 60 - 65 percent of maximal heart rate. After the warm-up and at the end of each training phase, the participants' heart rates were monitored. Finally, if the individual experienced pain, fainting, or shortness of breath, the training was promptly terminated
  Interventions: Procedure: Reflexology
- Reflexology (Experimental): This group consisted of twenty female patients suffering from hypertension who received the same drugs as group (A) as well as reflexology three times per week for eight weeks .
  Following four weeks of treatment (post-1) and additional four weeks of treatment (post-2) the post evaluation was used (post-2).Before and after the foot reflexology, blood pressure was checked twice. Around 20 minutes is spent on foot reflexology .
  Interventions: Procedure: Reflexology

INTERVENTIONS:
Procedure: Reflexology — Following four weeks of treatment (post-1) and additional four weeks of treatment (post-2) the post evaluation was used (post-2).Before and after the foot reflexology, blood pressure was checked twice. Around 20 minutes is spent on foot reflexology .
  Each patient in this study did 20 minutes of peddler aerobic training, with the first 5 minutes serving as a warm-up with intensity set at 60 - 65 percent of maximal heart rate, followed by another 10 minutes of peddler training with intensity gradually increased up to 70 - 75 percent, and the last 5 minutes serving as a cooling down with intensity set at 60 - 65 percent of maximal heart rate. After the warm-up and at the end of each training phase, the participants' heart rates were monitored. Finally, if the individual experienced pain, fainting, or shortness of breath, the training was promptly terminated as well as reflexology three times each week for eight weeks
  Other Names: Aerobic training

SUMMARY:
In Egypt, there is a dearth of understanding of the benefits of reflexology and aerobic exercise on hypertension patients' quality of life.

DETAILED DESCRIPTION:
The participated subjects were enrolled based on the inclusion and exclusion criteria , In this study, forty hypertensive female patients between 35 and 45 were divided to two equal groups (A and B). Twenty female patients in group (A) got medications and peddling training, while twenty female patients in group (B) had the exact treatment as group (A) as well as reflexology. Insomina severity index and a short form 36 quality of life questionnaire were used to assess the patients who took part in the study (ISI). They were assessed before and after the eight-week treatment program, which consisted of three sessions each week; following four weeks of treatment (post-1) and additional four weeks of treatment (post-2) the post evaluation was used (post-2).

ELIGIBILITY:
Inclusion Criteria:

1. Forty hypertensive patients aged 35 to 45 years of both sexes (men and women).
2. Clinical and medically, all of the participants were in good health.
3. The BMI ranged from 30 to 34.9 kg/m2 for all participants.

Exclusion Criteria:

1. Close Myocardial infarcts.
2. Heart block or complex ventricular arrhythmia
3. Cerebrovascular disease is a condition in which the blood vessels in the brain become inflamed.
4. Defects in vision or hearing.
5. Significant tightness in the lower limbs and/or a fixed deformity of lower limbs.
6. Balance or mentality-related neurological diseases (e.g. epilepsy).
7. Abnormalities of lower limb that may be congenital or acquired.

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Insomnia severity index | four weeks then four weeks( eight weeks)
  The Insomnia severity index is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia. The usual recall period is the "last month" and the dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, notice ability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem),
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe) The higher score is the worse outcome.
Short form 36 quality of life questionnaire (SF-36): | four weeks then four weeks( eight weeks)
  it is used for measuring health-related quality of life (HRQL) which consists of 36 questions (SF-36) (limitations on physical functioning because of health problems), it was done personal interviewing using Arabic version
Blood pressure measurements: | four weeks then four weeks( eight weeks)
  it consisted of systolic blood pressure which measures the pressure in arteries when heart beats and diastolic blood pressure which measures the pressure in arteries when heart rests between beats.

CONTACTS AND LOCATIONS:
Overall Officials: heba mousa, Principal Investigator — Cairo University
Locations (1):
- Heba Mousa, Cairo, Egypt

REFERENCES:
- [Background] Boutcher YN, Boutcher SH. Exercise intensity and hypertension: what's new? J Hum Hypertens. 2017 Mar;31(3):157-164. doi: 10.1038/jhh.2016.62. Epub 2016 Sep 8. PMID 27604656
- [Background] Gudsoorkar PS, Tobe SW. Changing concepts in hypertension management. J Hum Hypertens. 2017 Dec;31(12):763-767. doi: 10.1038/jhh.2017.57. Epub 2017 Jul 27. PMID 28748919